CLINICAL TRIAL: NCT05586529
Title: Effect of Preoperative High-dose Cholecalciferol in Prevention of Post-thyroidectomy Hypocalcaemia : A Randomized Controlled Trial
Brief Title: Effect of Preoperative High-dose Cholecalciferol in Prevention of Post-thyroidectomy Hypocalcaemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Mubashra Badar, Resident, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Thy 1 cpsp
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Hypocalcemia
Keywords: Cholecalciferol, post-operative hypocalcemia, thyroidectomy
MeSH Terms: conditions — Hypocalcemia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cholecalciferol group (Experimental): patients will recieve one dose of Vitamin D 200000 IU PO at the time of admission
  Interventions: Dietary Supplement: Cholecalciferol
- Control (No Intervention): Patients will not recieve any vitamin D before admission

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Cholecalciferol is vitamin D derivative and as our population already vit D deficient so post-operative hypocalcemia can be prevented.
  Other Names: Indrop-D
  Arms: Cholecalciferol group

SUMMARY:
Hypocalcaemia after thyroidectomy is observed with increasing frequency, often resulting in prolonged hospital stay with increased use of resources, delayed return to work and reduced quality of life. The administration of vitamin D is essential in the therapy of postoperative hypocalcaemia. What has not been examined so far is whether and how routine preoperative cholecalciferol prophylaxis can help to prevent postoperative hypocalcaemia

DETAILED DESCRIPTION:
Hypocalcemia following thyroid surgery is caused either due to parathyroid devascularization, stunning, or accidental removal of the parathyroid glandsMultiple risk factors have been identified which predispose patients to develop post-operative hypocalcemia. In light of the available evidence of prevalent vitamin D deficiency in the general population, and the observation of appearance of postthyroidectomy hypocalcemic symptoms at a much earlier stage than documented in previous literature, we postulate that a prophylactic vitamin D supplementation dose given in immediate preoperative period can significantly reduce acute symptomatic postoperative hypocalcemia in patients undergoing thyroid surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* Scheduled for TT
* Thyroid cancer treated with total thyroidectomy without lymph node dissection

Exclusion Criteria:

* Lack of written consent
* Thyroid cancer treated with TT and lymph node dissection
* Mediastinal goiter with need for sternotomy
* Medication with thiazide diuretics, digitalis or lithium therapy
* Previous neck operations or radiation
* Preexisting hyperparathyroidism
* Chronic kidney failure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative hypocalcemia | After 6 months
  The primary outcomes measure of this study was postoperative hypocalcemia based on either clinical symptoms or laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Mubashra Badar, Principal Investigator — Resident
Locations (1):
- Pak-Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Will publish this article and all the available darra will be available for researchers to view.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available once published.
Access Criteria: Any researcher who wants to buildup on this study